CLINICAL TRIAL: NCT03759444
Title: Stuck in Painful Time: Perception of Time by Individuals With Eating Disorders
Brief Title: Perception of Time by Individuals With Eating Disorders
Status: Completed | Type: Observational
Sponsor: Malgorzata Starzomska (Other)
Responsible Party: Sponsor-Investigator, Malgorzata Starzomska, Principal Investigator, Cardinal Stefan Wyszynski University
Organization: Cardinal Stefan Wyszynski University (Other)
Other Study IDs: PBF-31/16
Record Dates: First submitted 2018-11-20; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Feeding and Eating Disorders
Keywords: Perception of time; Eating disorders; Ego-syntonicity; Existential suffering; Psychotherapy
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with eating disorders: women with eating disorders (age: M = 26.88; SD = 5.82)
  The three measures applied in this group were: the Time Metaphors Questionnaire by Sobol-Kwapinska (2007), the Time Perspective Inventory by Zimbardo (1999), and the UWIST Mood Adjective Checklist (UMACL) by Matthews et al. (1990).
  Interventions: Other: Questionnaires
- healthy female controls.: healthy female controls (age: M = 24.27; SD = 6.49)
  The three measures applied in this group were: the Time Metaphors Questionnaire by Sobol-Kwapinska (2007), the Time Perspective Inventory by Zimbardo (1999), and the UWIST Mood Adjective Checklist (UMACL) by Matthews et al. (1990).
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The three questionnaires applied were: the Time Metaphors Questionnaire by Sobol-Kwapinska, the Time Perspective Inventory by Zimbardo, and the UWIST Mood Adjective Checklist (UMACL) by Matthews et al.

SUMMARY:
The objective of the study was to determine how patients with eating disorders perceive time, and in particular whether their experience of time differs from that of healthy individuals. Another goal was to examine the relationship between the mood of the subjects and their time perspective. The subjects were 30 women with eating disorders and 30 age-matched healthy female controls. The three measures applied were: the Time Metaphors Questionnaire by Sobol-Kwapinska, the Time Perspective Inventory by Zimbardo, and the UWIST Mood Adjective Checklist (UMACL) by Matthews et al.

DETAILED DESCRIPTION:
The objective of the study was to determine how individuals with eating disorders perceive time, and in particular whether their experience of time differs from that of healthy persons. Another aim was to investigate the relationship between the mood of the subjects and their time perception as well as determine a variable moderating that relationship.

First, it was expected that eating-disordered patients experience time as a rather aversive and unfriendly force marked with chaos and void, in contrast to healthy subjects, who were predicted to treat it as something more friendly, appreciating its subtleties and the significance of the moment (Hypothesis 1).

Moreover, it was expected that individuals with eating disorders would exhibit a more negative temporal orientation, whether past or present, as compared to healthy controls, who would reveal more positive past, present, or future orientations (Hypothesis 2).

Finally, it was predicted that eating disorders moderate the relationship between mood and time perception (Hypothesis 3).

The study encompassed 30 women with eating disorders (19 patients with anorexia nervosa and 11 patients with bulimia nervosa) and 30 age-matched normal healthy controls. The clinical group consisted of patients of the residential eating disorder therapeutic center "Drzewo zycia" in Malawa as well as some outpatient clinics in Poland; some of the patients were not being actively treated at the time of the study. The controls included psychology students from two Polish universities (the Cardinal Stefan Wyszynski University and the University of Finance and Management, both in Warsaw), as well as researchers and educators who volunteered for the study.

The three measures applied in the study were:

* The Time Metaphors Questionnaire by Sobol-Kwapinska;
* Time Perspective Inventory by Zimbardo (Zimbardo & Boyd, 1999; see also Zimbardo & Boyd, 2009);
* The UWIST Mood Adjective Checklist (UMACL) (Matthews at al.; see also Gorynska, 2005).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of eating disorders (anorexia nervosa or bulimia nervosa)
* Age between 18 and 40 years

Exclusion Criteria:

* diagnosis of other (except eating disorders) mental disorder
* Age below 18 years and above 40 years

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The clinical and control groups did not differ significantly in terms of age (t = 1.64, p = 0.100) or height (t = -0.54, p = 0.590). Obviously, significant differences were found in terms of weight and BMI (t = -2.93 and t = -3.03, p < 0.01, respectively): women with eating disorders were much lighter (M = 50.78, SD = 13.05) and had a much lower BMI (M = 18.3, SD = 4.49) than healthy controls (M = 60.43, SD = 12.48, and M = 21.62, SD = 3.98, respectively). The mean duration of eating disorder was 8.9 years (SD = 5.23).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
The Time Metaphors Questionnaire by Sobol-Kwapińska | 1.05.2014-30.06.2017
  The measure consists of 95 items formulated as metaphors describing ideas eliciting strong emotions. The subjects are asked to rate the items on a scale from 1 to 4, depending on the degree to which a given metaphor is consistent with their perception of time. The items are grouped into 3 scales reflecting positive attitudes to time: Friendly Time (subdivided into two subscales: Constructive Time and Pleasant Time), Significance of the Moment, and Subtle Time, as well as four scales covering negative attitudes to time: Hostile Time (with three subscales: Finiteness of Time, Bitter Time, and Confusion in Time), Rapid Passage of Time, Wild Time, and Empty Time. The questionnaire reveals satisfactory reliability and validity.
Time Perspective Inventory by Zimbardo | 1.05.2014-30.06.2017
  The measure consists of 56 items which the respondents rate on a 5-point scale ranging from 1 (very uncharacteristic of me) to 5 (very characteristic of me). The questionnaire tests 5 time perspectives: 1) Past-Negative, 2) Past-Positive, 3) Present-Hedonistic, 4) Present-Fatalistic, and 5) Future. The Polish version of this instrument has been reported to have both good reliability and validity.
Transcendental Future Time Perspective Inventory | 1.05.2014-30.06.2017
  This is a one-dimensional scale that consists of 10 items which the respondents rate on a 5-point scale ranging from 1 (very uncharacteristic of me) to 5 (very characteristic of me). It is used to assess individual attitudes and beliefs regarding the future, immediately following the imagined death of the physical body.
The UWIST Mood Adjective Checklist (UMACL) by Matthews et al. | 1.05.2014-30.06.2017
  The instrument measures mood understood as an affective experience of a duration of at least several minutes; its three scales are Tense Arousal, Energetic Arousal, and Hedonic Tone. The UMACL consists of a list of 29 adjectives which the respondents rate in terms of applicability to their current mood on a four-point scale from definitely yes to definitely not. The reliability and validity of the Polish adaptation has been confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Starzomska, dr, Principal Investigator — Cardinal Stefan Wyszynski University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gorynska E. UMACL Mood Adjective Checklist by G. Matthews, A.G. Chamberlain, D.M. Jones. Pracownia Testow Psychologicznych Polskiego Towarzystwa Psychologicznego, Warszawa, 2005.
- [Result] Matthews G, Jones DM, Chamberlain AG. Refining the measurement of mood: the UWIST Mood Adjective Checklist. British Journal of Psychology 81(1): 17-42, 1990.
- [Result] Sobol-Kwapinska M. TMQ Time Metaphor Questionnaire: Manual. Pracownia Testow Psychologicznych PTP, Warszawa, 2008.
- [Result] Zimbardo P G, Boyd J. The time paradox. PWN, Warszawa, 2009.
- [Result] Zimbardo P, Boyd J. Putting time in perspective: a valid, reliable individual differences metric. Journal of Personality and Social Psychology 77(6): 1271-1288, 1999.